CLINICAL TRIAL: NCT00702403
Title: A Multicenter Phase I/II Study of the Prophylactic Inhibition of BCR-ABL Tyrosine Kinase by Tasigna ® (Nilotinib) After Hematopoietic Cell Transplantation for Philadelphia Chromosome-Positive Leukemias.
Brief Title: Nilotinib and Imatinib Mesylate After Donor Stem Cell Transplant in Treating Patients With ALL or CML
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Paul Carpenter, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2223.00; NCI-2010-00402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Blastic Phase Chronic Myelogenous Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Chronic Phase Chronic Myelogenous Leukemia; Philadelphia Positive Adult Acute Lymphoblastic Leukemia; Philadelphia Positive Childhood Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia; Relapsing Chronic Myelogenous Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (prophylactic inhibition of BCR-ABL tyrosine kinase) (Experimental): Beginning after engraftment and blood count recovery (21 to 28 days after allogeneic stem cell transplant), patients with imatinib-sensitive leukemia receive imatinib mesylate PO QD until day 80 and then nilotinib PO BID on days 81-445. Patients with imatinib-resistant leukemia receive nilotinib PO BID beginning after engraftment and blood count recovery until day 445.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: nilotinib; Drug: imatinib mesylate; Other: pharmacological study

INTERVENTIONS:
Drug: nilotinib — Given PO
  Other Names: AMN 107; Tasigna
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial is studying the side effects and best way to give nilotinib when given alone or sequentially after imatinib mesylate after donor stem cell transplant in treating patients with acute lymphoblastic leukemia or chronic myelogenous leukemia. Nilotinib and imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of the administration of nilotinib between Day 81 and Day 365 after hematopoietic cell transplantation (HCT) in patients with Philadelphia chromosome positive (Ph+) leukemia.

SECONDARY OBJECTIVES:

I. To quantify the breakpoint cluster region (BCR)/Abelson murine leukemia (ABL) transcript load after HCT during tyrosine kinase inhibitor therapy in patients with Ph+ leukemia treated sequentially with imatinib (imatinib mesylate) and nilotinib from the time of engraftment.

II. To evaluate survival at 1 year in patients with Ph+ leukemia who received sequential imatinib and nilotinib from the time of engraftment.

III. To determine if imatinib can be co-administered with nilotinib for patients with rising levels of BCR/ABL on 2 consecutive occasions after HCT.

IV. To confirm that imatinib can be delivered at an average daily dose of 400 mg at least 85% of the time in the majority of adults during the first 80 days after HCT.

V. To determine whether nilotinib can be administered safely at a daily dose of at least 300 mg (175 mg/m^2 in children < 17 years) at least 70% of the time to patients with imatinib resistant Ph+ leukemia during the first 80 days after HCT.

VI. To determine treatment efficacy success at 1 year post-transplant as demonstrated by complete hematological remission, absence of Philadelphia chromosome, and not satisfying any of the criteria for treatment failure.

OUTLINE:

Beginning after engraftment and blood count recovery (21-28 days after allogeneic stem cell transplant), patients with imatinib-sensitive leukemia receive imatinib mesylate orally (PO) once daily (QD) until day 80 and then nilotinib PO twice daily (BID) on days 81-445. Patients with imatinib-resistant leukemia receive nilotinib PO BID beginning after engraftment and blood count recovery until day 445.

Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Body surface area >= 1 m^2
* Allogeneic HCT
* Acute lymphocytic leukemia (ALL) or chronic myelogenous leukemia (CML) characterized by the p190 and/or p210 BCR/ABL gene rearrangement
* CML in accelerated phase, blast crisis, or blast crisis remission as defined by World Health Organization (WHO) criteria
* CML in chronic phase if patient age =< 17 years or a patient of any age with CML in second chronic phase or beyond
* Patients with minimal residual disease (MRD) that is not declining in response to tyrosine kinase inhibitor therapy must be screened for the T315I and other mutations
* An appropriately matched related or unrelated donor
* Signed informed consent
* Patient must have a life expectancy of at least 2 months
* Stated willingness of the patient to comply with study procedures and reporting requirements
* Creatinine =< 2.0 x upper limit normal (ULN)
* Platelets > 20 x 10^9 /L
* Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN, conjugated bilirubin < 3 x ULN
* Serum potassium phosphorus, magnesium, and calcium >= lower limit normal (LLN) or correctable with supplements prior to first dose of study drug; calcium levels may be corrected for hypoalbuminemia
* Serum amylase and lipase < 1.5 x ULN
* Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing; postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential; male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Careful rationalization with a view to discontinuing or considering alternatives to any concomitant medications that have potential to prolong the QT interval

Exclusion Criteria:

* Autologous transplant
* Non-myeloablative transplant
* Patient age > 17 years with CML in first chronic phase
* Aberrant antigen expression on marrow leukemic blasts >= 5% by multidimensional flow cytometric assay immediately before conditioning (CML patients in chronic phase exempt from flow cytometry screening)
* Ph+ ALL without complete cytogenetic remission immediately before conditioning
* Known T315I mutation
* Hypersensitivity to Gleevec or Tasigna
* Patients who are Tasigna-resistant or intolerant
* Central nervous system (CNS) involvement with leukemia at baseline (pre-imatinib therapy); CML chronic phase (CP), accelerated phase (AP) patients exempt from CNS involvement screening
* Female patients who are pregnant, breast-feeding, or of childbearing potential without a negative serum pregnancy test at screening; male or female patients of childbearing potential unwilling to use effective contraceptive precautions throughout the trial; post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
* Life expectancy severely limited by diseases other than leukemia
* Myocardial infarction within one year prior to starting nilotinib
* Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, unstable angina)
* Absolute neutrophil count (ANC) less than 1500 per microliter at study entry despite the use of filgrastim (G-CSF)
* Impaired cardiac function, including any one of the following:

  * Complete left bundle branch block or bifascicular block (right bundle branch block plus left anterior hemiblock) or use of ventricular-paced pacemaker
  * Congenital long QT syndrome or a family history of long QT syndrome
  * History of or presence of significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats per minute)
* Corrected QT interval (QTc) > 450 milliseconds on screening electrocardiogram (ECG); if QTc > 450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient rescreened for QTc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-08-14 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Carpenter, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (5):
  - Stanford University Hospitals and Clinics, Stanford, California
  - H Lee Moffitt Cancer Center and Research Institute Phase 2 Consortium, Tampa, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Oregon Health and Science University, Portland, Oregon
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Nilotinib Relapse Prophylaxis: Beginning after engraftment and blood count recovery (21 to 28 days after allogeneic stem cell transplant), patients with imatinib-sensitive leukemia receive imatinib mesylate PO QD until day 80 and then nilotinib PO BID on days 81-445. Patients with imatinib-resistant leukemia receive nilotinib PO BID beginning after engraftment and blood count recovery until day 445. Treatment continues in the absence of disease progression or unacceptable toxicity.
Period: From Consent to Engraftment
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
Started | 57 (57 agreed to participate and completed informed consent (= the 1st "intention to treat" population))
Ineligible for Study Drug | 17
Completed | 40 (40 of 57 originally consented subjects remained eligible at engraftment (= the 2nd ITT population))
Not Completed | 17
Not completed — Progressive leukemia | 6
Not completed — Critically ill | 2
Not completed — Corrected QT interval (QTc) >450 msec | 2
Not completed — Myocardial infarction | 1
Not completed — ANC<1500, plts<20K or hyperbilirubinemia | 4
Not completed — Miscellaneous (unanticipated) other | 2
Period: From Engraftment to Study Completion
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
Started | 40
Patient Drop-outs | 27
Completed | 13
Not Completed | 27
Not completed — Failed pre-1st dose criteria | 11
Not completed — Relapse (1 Central Nervous System, 3 BM) | 4
Not completed — Non-compliance | 2
Not completed — Adenocarcinoma | 1
Not completed — Liver GVHD | 1
Not completed — Suicide | 1
Not completed — Acute respiratory distress syndrome | 1
Not completed — Dyspnea (unrelated to nilotinib) | 1
Not completed — Toxicity attributed to Nilotinib | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 42.5 [11 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 33
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Safety Failure
Description: Safety and tolerability of nilotinib therapy in patients with imatinib-sensitive leukemia graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version 4.0. Treatment safety failure is defined for a patient with imatinib sensitive Ph+ leukemia as the inability to be able to deliver at least 400 milligrams per day of nilotinib in adults, and 230 milligrams/m2 per day in children, for at least 85% of the time interval between 81 and 365 days after transplant. The overall study will be considered successful if nilotinib is deliverable to more than 75% of the study participants at this minimum specified dose intensity.
Time Frame: Up to 365 days post-transplant
Population: Critical to note are two "intention-to-treat" populations: the 1st (N=57) at time of consent, evolved into the second ITT population (N=40), because 17 subjects lost eligibility to begin relapse prophylaxis at engraftment. A 2nd wave of discontinuations occurred at or after Day 81 when all patients were to be switched from imatinib to nilotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
Number analyzed (Participants) | 40
Participants | 13

2. Secondary Outcome: The Proportion of Patients at 1 Year With Treatment Efficacy Success
Description: To be considered a treatment efficacy success at 1 year posttransplant, the patient's bone marrow must demonstrate complete hematological remission, absence of Philadelphia chromosomes, and not satisfy any of the criteria for treatment failure (>/= 1% aberrantly expressing marrow blasts by multiparameter flow cytometry, >5% BCR/ABL in marrow by fluorescent in situ hybridization, or >1 log rise in peripheral blood BCR/ABL by quantitative polymerase chain reaction (PCR) since day 80).
Time Frame: Up to 1 year
Population: The analysis population was considered in two ways: first the number of treatment success in the entire cohort (by "intention to treat"), and second the number of treatment successes among only those patients who did not die before 1 year from non-relapse mortality.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Prophylactic Inhibition of BCR-ABL Tyrosine Kinase): Beginning after engraftment and blood count recovery (21 to 28 days after allogeneic stem cell transplant), patients with imatinib-sensitive leukemia receive imatinib mesylate PO once daily until day 80 and then nilotinib PO twice daily on days 81-445. Patients with imatinib-resistant leukemia receive nilotinib PO twice daily beginning after engraftment and blood count recovery until day 445. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Prophylactic Inhibition of BCR-ABL Tyrosine Kinase)
Number analyzed (Participants) | 40
Participants
  By intention to treat | 29
  Excluding early non-relapse deaths: number analyzed (Participants) | 34
  Excluding early non-relapse deaths | 29

3. Secondary Outcome: Survival
Description: The proportion of study participants alive at 1, 2 and 3 years
Time Frame: Up to 3 years
Population: Overall Survival (complete follow-up is available out to three years for all patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Prophylactic Inhibition of BCR-ABL Tyrosine Kinase)
Number analyzed (Participants) | 40
Participants
  Overall Survival at 1 year | 31
  Overal Survival at 2 years | 28
  Overall Survival at 3 years | 28

4. Secondary Outcome: Patients Alive With Out Relapse
Description: The proportion of study participants alive and without hematologic, cytogenetic or molecular evidence of BCR/ABL-positive leukemia at 1 year
Time Frame: Up to 1 year
Population: Proportion alive without relapse among the total number of patients with minimal residual disease follow-up data
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm Nilotinib Relapse Prophylaxis: Beginning after engraftment and blood counts recover (21 to 28 days after allogeneic stem cell transplant), patients with imatinib-sensitive leukemia receive imatinib mesylate PO once daily until day 80 and then nilotinib PO twice daily on days 81-445. Patients with imatinib-resistant leukemia receive nilotinib PO twice daily beginning after engraftment and blood counts recover until day 445. Treatment continues in the absence of disease progression or unacceptable toxicity.
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
Number analyzed (Participants) | 40
Participants | 29

5. Secondary Outcome: Relapse
Description: The proportion of patients with hematologic, cytogenetic or molecular relapse of BCR/ABL-positive leukemia
Time Frame: 1 and 3 years
Population: Proportion of patients with hematologic, cytogenetic or molecular relapse of BCR/ABL-positive leukemia among those who did not die from non-relapse causes during the first year, and first 3-years after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Prophylactic Inhibition of BCR-ABL Tyrosine Kinase)
Number analyzed (Participants) | 40
Participants
  Proportion with relapse at 1 year | 5
  Proportion with relapse at 3 years | 6

ADVERSE EVENTS:
Time Frame: Adverse Events: Conditioning through Day 100; Severe Adverse Events Conditioning >Day 100
Arm/Group | Single Arm Nilotinib Relapse Prophylaxis
All-Cause Mortality (participants affected / at risk) | 9/40
Serious Adverse Events (participants affected / at risk) | 20/40
Other Adverse Events (participants affected / at risk) | 31/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Nilotinib Relapse Prophylaxis (N=40)
Acute acalculous cholecystitis (Hepatobiliary disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 1
Transaminitis (Hepatobiliary disorders) | 1
Pseudomonas bacteremia (Infections and infestations) | 1
Gram negative rod bacteremia with possible urosepsis (Infections and infestations) | 1
Cytomegalovirus reactivation (Infections and infestations) | 1
Fever/URI (Infections and infestations) | 2
Staph Aureus Bacteremia (Infections and infestations) | 1
Alpha-hemolytic Streptococcus (Infections and infestations) | 1
Staph haemolyticus (Infections and infestations) | 1
Gram-negative Bacteremia and Septic emboli (Infections and infestations) | 1
Nodular pneumonia (Infections and infestations) | 1
Bacterial pneumonia (Infections and infestations) | 1
Acute lobular pneumonia with sepsis (Infections and infestations) | 1
Haemophilus Influenza-Rhinovirus (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pericardial effusion (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1
Malignant hypertension (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Yeast esophagitis-Odynophagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Abdominal Cramping (Gastrointestinal disorders) | 1
Headache (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Transaminitis (Gastrointestinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Non-specific interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Altered mental status (Psychiatric disorders) | 1
Acute encephalopathy (Psychiatric disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Death, NOS (General disorders) | 1
Generalized weakness/fatiuge (General disorders) | 1
Multiorgan failure (General disorders) | 1
Hemorrhagic cystitis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Nilotinib Relapse Prophylaxis (N=40)
Klebsiella pneumonia pyelonephritis and positive urine culture (Infections and infestations) | 1
Vancomycin resistant enterococcus and positive urine culture (Infections and infestations) | 1
Bacteremia enterococcus faecalis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
CMV Reactivation (Infections and infestations) | 7
Coagulase-negative staph (Infections and infestations) | 3
CMV Enteritis (Infections and infestations) | 1
Candidal esophagitis (Infections and infestations) | 1
BK Virus (Infections and infestations) | 2
Klebsiella and E.Coli and Positive Urine Culture (Infections and infestations) | 1
S. epidermidis bacteremia (Infections and infestations) | 1
Pseudomonas maltophilia Bacteremia (Infections and infestations) | 1
GPC Bacteremia (Infections and infestations) | 1
Multiorganism sepsis (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 19
Anemia (Blood and lymphatic system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 7
Lymphocytopenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 6
INR Increased (Blood and lymphatic system disorders) | 1
Cytopenia (Blood and lymphatic system disorders) | 2
Elevated Serum AST/ALT (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Anorexia/Nausea (Metabolism and nutrition disorders) | 1
Increased Bilirubin (Metabolism and nutrition disorders) | 1
Increased Alkaline Phosphate (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Increased creatinine-renal insufficiency (Metabolism and nutrition disorders) | 1
Increased Lipase (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 1
Localized Edema (General disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1
Renal Disease (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Delerium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes